CLINICAL TRIAL: NCT05370339
Title: Assessment of Sleep and Sleep Disruptors in Adolescents With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 21-4311
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes; Insufficient Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents: Adolescents with type 1 diabetes between the ages of 11 and 17 years.

SUMMARY:
The goal of this study is to identify causes of insufficient sleep and sleep disruptors in adolescents with type 1 diabetes. For this study, adolescents will wear an actigraphy watch and complete sleep diaries for seven days. On completion of the seven days, they will complete several questionnaires regarding sleep, fear of hypoglycemia, and anxiety and depression. A subset of participants will additionally complete a qualitative interview session to obtain a deeper understanding of sleep disruptors and barriers and facilitators to improving sleep health.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T1D at least 3 months
* Receive clinical care at the Barbara Davis Center

Exclusion Criteria:

* Have an active underlying sleep disorder, such as narcolepsy, insomnia, or untreated sleep apnea
* Participation in an interventional research protocol
* Unable to complete study procedures

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents with type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Number of nocturnal awakenings per week | One week per participant
  We will identify the number of nocturnal awakenings per week for comparison of those with insufficient sleep identified by actigraphy watch to those with sufficient sleep.
Assessment of facilitators and barriers to good sleep quality and duration | One week per participant
  Qualitative interviews will be conducted and analyzed for themes to identify causes of sleep disruptions and any potential barriers or facilitators to improving sleep health.

SECONDARY OUTCOMES:
Identification of common causes of sleep disruptors in adolescents with type 1 diabetes | One week per participant
  Sleep diaries will be used to determine common causes of sleep disruptors in adolescents with type 1 diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No